CLINICAL TRIAL: NCT02023567
Title: The Establishment of the Objective Diagnostic Markers and Personalized Medical Intervention in Patients With Major Depressive Disorders (MDD)
Brief Title: Objective Diagnostic Markers and Personalized Intervention in MDD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Capital Medical University (Other); Peking Union Medical College Hospital (Other); Tianjin Medical University General Hospital (Other); Tianjin Anding Hospital (Other); The First Hospital of Hebei Medical University (Other); First Hospital of China Medical University (Other); Dalian Seventh People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Xin Yu, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013CB531305
Record Dates: First submitted 2013-12-15; First posted 2013-12-30 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDD group (Experimental): Drugs: SSRIs fluoxertine hydrochloride (20- 60m/day),paroxetine hydrochloride (20- 60m/day),sertraline hydrochloride (50- 200m/day),citalopram (20-60m/day), escitalopram (10-20mg/day),fluvoxamine (50-300mg/day)
  Interventions: Drug: SSRIs
- Healthy controls (No Intervention): This group just receive baseline evaluation and did not receive any intervention.

INTERVENTIONS:
Drug: SSRIs — fluoxertine hydrochloride 20-60mg/day, paroxetine hydrochloride 20-60mg/day, sertraline hydrochloride 50-200mg/day, citalopram 20-60mg/day, escitalopram 10-20mg/day, fluvoxamine 50-300mg/day
  Other Names: selective serotonin reuptake inhibitors
  Arms: MDD group

SUMMARY:
Major depressive disorder (MDD) is one of the most common psychiatric disorders, with high recurrence rate, suicide rate and disability rate. It's reported that the global burden caused by MDD will be up to the second rank among all the disease burdens by 2020. China is also confronted with the daunting challenges against MDD. It's assessed that the monthly incidence of MDD is 6.1%, non-hospitalizing rate reaches up to 92% and the non-treatment rate is approximate 95%. However, to date, the pathogenesis of MDD is obscure and the current therapies don't work well. Therefore, it's urgent and critical to elucidate the pathogenesis of MDD, to develop early diagnostic criteria and effective intervention in MDD. Considering the diversity of weights on genetic factor and environmental factor in MDD, in this project, the investigators aim firstly to explore the effect of "genetic-environmental interaction"on the pathogeny of MDD for classifying MDD into "genetic type", "environmental type" and "others" based on a case-control study. We next conduct the neurobiological, neurocognitive and psycho-behavioral assessments among MDD, schizophrenia and healthy groups to screen the salient endophenotypes for establishing the diagnostic models of MDD . The investigators further analyse the changes of these indicators after 8 weeks'medication to select the potential predictors for therapeutic evaluations and interventional options in MDD patients. Finally, the investigators continue a 2-year follow-up study to test and verify the predictors of prognosis in MDD patients.

ELIGIBILITY:
1. For MDD group:

   Inclusion criteria:
   * Age between 18-55, male or female;
   * The diagnosis of MDD consistent with DSM-IV (M.I.N.I)
   * First-episode or relapsed;
   * Certain ability of reading and writing to complete the questionnaire survey and psychological assessment.
   * All participants provide written confirmation of informed consent prior to engaging the study protocol.

   Exclusion criteria:
   * Current psychopathology or a history of neurologic conditions, including alcohol/substances dependence, the diagnosis of cognition impairment;
   * Severe somatic diseases, such as severe cardio-cerebral vascular diseases, respiratory diseases, liver diseases, kidney diseases, or malignant tumors;
   * Not signed the informed consent;
   * Been engaging other studies.
2. For Healthy control group

Inclusion criteria:

* age between 18 and 55 years at the time of enrollment;
* providing written confirmation of informed consent prior to engaging the study.

Exclusion criteria:

* lifetime or current diagnosis of any mental diseases;
* severe somatic diseases, such as severe cardio-cerebral vascular diseases, respiratory diseases, liver diseases, kidney diseases, or malignant tumors;
* not signed the informed consent;
* been engaging other studies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2400 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The changes of HAMD total score at 8 weeks from baseline | week 0,2,4,8
  The scores are assessed at 0,2,4,8 weeks since the medication begins for MDD group

SECONDARY OUTCOMES:
The changes of HAMA total score at 8 weeks from baseline | week 0,2,4,8
  The scores are assessment at 0,2,4,8 weeks since the medication begins for MDD group
The change of CGI score at 8 weeks from baseline | week 0,2,4,8
  The scores are assessment at 0,2,4,8 weeks since the medication begins for MDD group
The prognosis after the intervention | Up to 2 years
Number of participants with serious and non-serious adverse events | Up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, MD, Principal Investigator — Peking University Sixth Hospital
Locations (9):
- China (9):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Hebei Medical University First Hospital, Shijiazhuang, Hebei
  - Dalian Seventh People's Hospital, Dalian, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided
After enrollment completion,we will decided whether share data or not.

REFERENCES:
- [Derived] Cui F, Liu Q, Lv X, Tian H, Wei J, Zhang K, Zhu G, Chen Q, Wang G, Wang X, Zhang N, Huang Y, Si T, Yu X. Effect of childhood trauma on cognitive function in individuals with major depressive disorder and healthy controls. J Affect Disord. 2025 Feb 15;371:196-204. doi: 10.1016/j.jad.2024.10.059. Epub 2024 Oct 19. PMID 39433132
- [Derived] Lin J, Li JT, Kong L, Liu Q, Lv X, Wang G, Wei J, Zhu G, Chen Q, Tian H, Zhang K, Wang X, Zhang N, Yu X, Si T, Su YA. Proinflammatory phenotype in major depressive disorder with adulthood adversity: In line with social signal transduction theory of depression. J Affect Disord. 2023 Nov 15;341:275-282. doi: 10.1016/j.jad.2023.08.104. Epub 2023 Aug 30. PMID 37657624
- [Derived] Lin J, Su Y, Lv X, Liu Q, Wang G, Wei J, Zhu G, Chen Q, Tian H, Zhang K, Wang X, Zhang N, Yan H, Wang Y, Yu X, Si T. Childhood adversity, adulthood adversity and suicidal ideation in Chinese patients with major depressive disorder: in line with stress sensitization. Eur Arch Psychiatry Clin Neurosci. 2022 Aug;272(5):887-896. doi: 10.1007/s00406-021-01375-4. Epub 2022 Jan 5. PMID 34985583
- [Derived] Cui F, Liu Q, Lv X, Leonhart R, Tian H, Wei J, Zhang K, Zhu G, Chen Q, Wang G, Wang X, Zhang N, Huang Y, Si T, Yu X. Severe sleep disturbance is associated with executive function impairment in patients with first-episode, treatment-naive major depressive disorders. BMC Psychiatry. 2021 Apr 19;21(1):198. doi: 10.1186/s12888-021-03194-2. PMID 33874911
- [Derived] Lin J, Su Y, Lv X, Liu Q, Wang G, Wei J, Zhu G, Chen Q, Tian H, Zhang K, Wang X, Zhang N, Wang Y, Yu X, Si T. Perceived stressfulness mediates the effects of subjective social support and negative coping style on suicide risk in Chinese patients with major depressive disorder. J Affect Disord. 2020 Mar 15;265:32-38. doi: 10.1016/j.jad.2020.01.026. Epub 2020 Jan 10. PMID 31959583
- [Derived] Lin JY, Huang Y, Su YA, Yu X, Lyu XZ, Liu Q, Si TM. Association between Perceived Stressfulness of Stressful Life Events and the Suicidal Risk in Chinese Patients with Major Depressive Disorder. Chin Med J (Engl). 2018 Apr 20;131(8):912-919. doi: 10.4103/0366-6999.229898. PMID 29664050
- [Derived] Lv X, Si T, Wang G, Wang H, Liu Q, Hu C, Wang J, Su Y, Huang Y, Jiang H, Yu X. The establishment of the objective diagnostic markers and personalized medical intervention in patients with major depressive disorder: rationale and protocol. BMC Psychiatry. 2016 Jul 15;16:240. doi: 10.1186/s12888-016-0953-z. PMID 27422150